CLINICAL TRIAL: NCT07267845
Title: A Randomised, Double-Blind, Placebo-Controlled Study on the Effects of Alpha-Glycerophosphocholine (α-GPC) on Cognitive Function and Sports Performance in Adults
Brief Title: The Effect of α-GPC on Cognitive Function and Sports Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Nutrabuilding Bio-tech Co., Ltd. (Other)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NNB2025HCS-AFCRO-199
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Alpha-Glycerophosphocholine; α-GPC; cognitive function; sports performance; Dietary Supplement; safety
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement: 315 mg α-GPC (Experimental)
  Interventions: Dietary Supplement: Alpha-Glycerophosphocholine（α-GPC）
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Microcrystalline Cellulose (placebo)

INTERVENTIONS:
Dietary Supplement: Alpha-Glycerophosphocholine（α-GPC） — Participants will oral one capsule containing 350 mg of GeniusPure® (containing 315 mg of pure α-GPC) daily before breakfast for 6 weeks.
  Arms: Dietary Supplement: 315 mg α-GPC
Dietary Supplement: Microcrystalline Cellulose (placebo) — Participants will oral one capsule containing 350 mg of microcrystalline cellulose (MCC) daily before breakfast for 6 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to find out whether daily supplementation with Alpha-Glycerophosphocholine (α-GPC) can improve cognitive function and sports performance in healthy adults. It will also assess the safety and tolerability of α-GPC when taken over a 6-week period.

The main questions this study aims to answer are:

Does taking α-GPC every day improve cognitive performance on tests such as the Stroop Test, Go/No-go Test, Sustained Attention to Response Task (SART), and Digit-Symbol Substitution Test (DSST)? Does α-GPC enhance upper and lower body sports performance? Does α-GPC positively affect perceived mood, energy, and motivation? Is α-GPC safe and well tolerated compared to a placebo? Researchers will compare α-GPC (350 mg per day) to a placebo (an inactive substance that looks the same) in a randomized, double-blind study. Neither the participants nor the researchers will know who receives α-GPC or the placebo.

Participants will:

Be randomly assigned to take either α-GPC or placebo capsules once daily for 6 weeks Attend 3 study visits over an 8-week period at Atlantia Clinical Trials in Cork, Ireland Complete cognitive and physical performance tests both acutely (shortly after a single dose) and after 6 weeks of daily use Have their vital signs, body weight, and any adverse events monitored throughout the study Record their diet and well-being during the study period This study will include 80 healthy adults aged 25-55 years who regularly engage in physical activity. The results will help determine whether α-GPC has benefits for brain function and physical performance, and whether it is safe for long-term use.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be in good health as determined by the investigator.
* Age between 25 and 55 years (inclusive).
* Body Mass Index of 18.5-32.0 kg/m2 (inclusive).
* Body weight of at least 54 kilograms.
* Muscle strengthening activities 2-3 time per week or participation in recreational or local level moderate intensity activity for at least 2 years.
* Normotensive (resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg).
* Willing to duplicate their previous 24-hr diet, refrain from alcohol and caffeine for 24-hr prior to each visit, refrain from exercise 48-hr prior to each visit.
* Refrain from consuming beef liver, chicken liver, eggs, fish, wheat germ and soybeans, butter beans 24-hrs prior to Visit 2 and Visit 3.

Exclusion Criteria:

* Highly trained or competitive athletes.
* Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
* Female participants who are currently breastfeeding.
* Female participants who are planning to become pregnant during the study period.
* Female participants who test positive on a pregnancy test at screening or prior to first administration of the study product.
* Participants with history of drug and/or alcohol abuse at the time of enrolment. (Drinks more than nationally recommended units per week (>11 units for women; >17 units for men); alcohol/substance abuse disorder).
* Caffeine intake of three or more cups of coffee or equivalent (>400 mg) per day.
* Current smokers or users of any nicotine products in the past 4-weeks.
* Has food allergies or other issues with foods that would preclude intake of the Study Products.
* Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer.
* Diagnosed, uncontrolled psychiatric disorder.
* Hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Prior gastrointestinal bypass surgery (excluding appendectomy).
* Gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism.
* Chronic inflammatory condition or disease.
* History of severe or chronic musculoskeletal pain or injury.
* History of diabetes, asthma, gout, fibromyalgia or clinical diagnosis of IBS/IBD.
* Current or recent use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results as judged by the investigator.
* Use CNS stimulants or anxiety or ADHD medication.
* Use corticosteroids (oral, subcutaneous, intramuscular, or transdermal only).
* Use testosterone replacement therapy (ingestion, injection, or transdermal).
* Current or recent use of prohibited nutritional or non-nutritional supplements that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results as judged by the investigator.
* Use creatine, BCAA, HMB, betaine, beta-alanine, in the past 2 weeks.
* Use choline supplements (e.g. choline bitartrate, phosphatidylcholine, citicholine) in the past 4 weeks.
* Use omega-3, ginkgo biloba, ginseng, L-theanine, Lion's Mane, ashwagandha in the past 4 weeks.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
* Participants may be participating in other clinical studies.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance - Stroop Test-Stroop total score | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the stroop total score change (Δ) of from Day 1 to Day 42 in the α-GPC group compared to placebo on Stroop Test.

SECONDARY OUTCOMES:
Cognitive Performance - Stroop Test - Stroop accuracy (%) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the stroop accuracy (%) change (Δ) of from Day 1 to Day 42 in the α-GPC group compared to placebo on Stroop Test.
Cognitive Performance - Stroop Test - Stroop time per score (s) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the stroop time per score (s) change (Δ) of from Day 1 to Day 42 in the α-GPC group compared to placebo on Stroop Test.
Cognitive performance - Digit-Symbol Substitution Test (DSST) - Number of Correct Symbols (N) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the Number of Correct Symbols (N) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Digit-Symbol Substitution Test (DSST) - Total Correct Score | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the Total Correct Score change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Digit-Symbol Substitution Test (DSST) - Accuracy (%) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the Accuracy (%) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Digit-Symbol Substitution Test (DSST) - Time per Correct Response (s/item) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test the Time per Correct Response (s/item) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test - Correct responses (N) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Go/No-Go - Correct responses (N) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test - Errors of omissions (%) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Go/No-Go - Errors of omissions (%) change (Δ) from Day 1 to Day 42 effect in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test - Errors of commission (%) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Go/No-Go - Errors of commission (%) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test - Correct rejections (N) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Go/No-Go - Correct rejections (N) change (Δ) from Day 1 to Day 42 effect in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test - Mean response times (mins) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Go/No-Go - Mean response times (mins) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test - Reaction time (mins) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Reaction time (mins) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive performance - Go/No-go Test- Reaction time variability (RTV) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the Reaction time variability (RTV) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive Performance - Sustained Attention to Response Task (SART) - Total Commission Errors (N) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test total commission errors (N) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive Performance - Sustained Attention to Response Task (SART) - Omission Errors (N) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test omission errors (N) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive Performance - Sustained Attention to Response Task (SART) - Reaction Time (Mean RT) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test reaction time (Mean RT) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo.
Cognitive Performance - Sustained Attention to Response Task (SART) - Reaction Time Variability (RTV) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）
  Test reaction time variability (RTV) change (Δ) from Day 1 to Day 42 effect in the α-GPC group compared to placebo on.
Upper Body Power - Average power (W) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  The average power (W) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to the Placebo group will be assessed by Ballistic Smith Machine Bench Press.
Upper Body Power - Peak power production (W) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  The peak power production (W) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to the Placebo group will be assessed by Ballistic Smith Machine Bench Press.
Upper Body Power - Peak Velocity (m/s) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  The peak velocity (m/s) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to the Placebo group will be assessed by Ballistic Smith Machine Bench Press.
Upper Body Power - Peak force production (N) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  The peak force production (N) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to the Placebo group will be assessed by Ballistic Smith Machine Bench Press.
Lower Body Power - Average power (W) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the average power (W) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo on Vertical Jump for Lower Body Power (Tendo).
Lower Body Power - Peak power production (W) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the peak power production (W) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo on Vertical Jump for Lower Body Power (Tendo).
Lower Body Power - Peak Velocity (m/s) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the peak Velocity (m/s) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo on Vertical Jump for Lower Body Power (Tendo).
Lower Body Power - Peak force production (N) | Assessed 90 minutes after ingestion of assigned test product during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Test the peak force production (N) change (Δ) from Day 1 to Day 42 in the α-GPC group compared to placebo on Vertical Jump for Lower Body Power (Tendo).
Perceived mood assessment | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Perceived mood assessed using the Visual Analog Scale (VAS), a 0-100 scale where 0 indicates 'worst mood imaginable' and 100 indicates 'best mood imaginable.' Higher scores represent better perceived mood.
Perceived motivation assessment | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Perceived motivation assessed using the Visual Analog Scale (VAS), with a range of 0-100 where 0 indicates 'no motivation' and 100 indicates 'maximum motivation.' Higher scores represent better perceived motivation.
Perceived energy assessment | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Perceived energy assessed using the VAS, with a range of 0-100 where 0 indicates 'no energy' and 100 indicates 'maximum energy.' Higher scores represent better perceived energy.

OTHER OUTCOMES:
Heart Rate Measurement | Assessed at 0(before ingestion of assigned test product ), 60 and 190 min(after ingestion product) during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Accurately measure heart rate using a dedicated heart rate monitor.
Blood Pressure Measurement (Systolic and Diastolic) | Assessed at 0(before ingestion of assigned test product ), 60 and 190 min(after ingestion product) during baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Blood pressure measured using an automated sphygmomanometer. Both systolic and diastolic pressures will be assessed.
Dietary Energy Intake | During baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  24-Hour Dietary Intake using 24-hour recall approach.Dietary calorie intake(kcal) were evaluated.
Dietary macronutrient intake | During baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  24-Hour Dietary Intake using 24-hour recall approach. Dietary macronutrient intake(g) were evaluated.
Temperature | During baseline（visit 2, week 1, day1） and end of the study（visit 3, week 6, day42）.
  Forehead temperature was measured using an electronic thermometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, Cork, County Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scientists help craft gene testing law. Science. 1996 Mar 1;271(5253):1235, 1237. No abstract available. PMID 11644786
- [Result] Gatti G, Barzaghi N, Acuto G, Abbiati G, Fossati T, Perucca E. A comparative study of free plasma choline levels following intramuscular administration of L-alpha-glycerylphosphorylcholine and citicoline in normal volunteers. Int J Clin Pharmacol Ther Toxicol. 1992 Sep;30(9):331-5. PMID 1428296
- [Result] Yamashita S, Kawada N, Wang W, Susaki K, Takeda Y, Kimura M, Iwama Y, Miura Y, Sugano M, Matsuoka R. Effects of egg yolk choline intake on cognitive functions and plasma choline levels in healthy middle-aged and older Japanese: a randomized double-blinded placebo-controlled parallel-group study. Lipids Health Dis. 2023 Jun 20;22(1):75. doi: 10.1186/s12944-023-01844-w. PMID 37340479